CLINICAL TRIAL: NCT05260892
Title: Incisors Single-Unit Rehabilitation With Narrow GM Implants: Observational Prospective Study
Brief Title: Incisors Single-Unit Rehabilitation With Narrow GM Implants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Other Study IDs: CS.O.004
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Edentulous Alveolar Ridge
Keywords: dental implants; oral rehabilitation; extra narrow implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Narrow GM: Patients presenting at least onde edentulous site rehabilitated with Narrow GM implant
  Interventions: Device: Narrow GM implants

INTERVENTIONS:
Device: Narrow GM implants — Rehabilitation of superior lateral incisors or inferior central and lateral incisors with narrow implants supporting single unit or partial prostheses

SUMMARY:
The Narrow GM Implants were designed for oral functional rehabilitation using dental implants, allowing for treatment of patients with different bone qualities in the region of lateral incisors in the maxilla or the region of lateral and central incisors in the mandible.

The objective of the study is to confirm the long-term safety and clinical performance of implants and abutments of the Narrow GM System in a daily dental practice setting, by means of a prospective collection of clinical data in an observational study using these devices.

Devices will be used according to standard routine in daily practice, according to all indications as specified by the manufacturer in the instructions for use (IFU).

55 patients (needed to obtain a sample size of 55 implants) will be followed for 36 months and monitored for Adverse Events by the Investigators until the last protocol-related procedure of a patient is completed.

DETAILED DESCRIPTION:
The study protocol was reviewed and approved by an Ethics Committee (CE) in Brazil.

The Narrow GM Implants were designed for oral functional rehabilitation using dental implants, allowing for treatment of patients with different bone qualities in the region of lateral incisors in the maxilla or the region of lateral and central incisors in the mandible.

The objective of the study is to confirm the long-term safety and clinical performance of implants and abutments of the Narrow GM System in a daily dental practice setting, by means of a prospective collection of clinical data in an observational study using these devices. Additionally, from the collected data, the study aims to identify previously unknown side-effects and monitor the known side-effects and contraindications stated on the Instruction for Use (IFU), identify and analyze emerging risks on the basis of factual evidence and ensure the continued acceptability of the benefit-risk ratio with the intent to verify that the intended purpose is correct for all JJGC products involved in the procedure that get in contact with the patient.

The sample will be prospectively selected and will consist of 55 patients, with at least one edentulous site in the region of lateral incisors in the maxilla and/or lateral and central incisors in the mandible, presenting natural adjacent and opposing tooth, and who are qualified for rehabilitation with narrow implants and single-unit fixed prostheses. Informed consent in writing will be obtained from each patient participating in the study prior to any study-related procedure.

GM Narrow implants will be placed under local anesthesia by guided or conventional surgery - as chosen by the surgeon - and with adequate bone bed preparation, as recommended by the manufacturer. Multiple implants can be placed in the same patient, as indicated. Implants must be installed 2mm infra-bony.

Data concerning the studied variables will be collected following the procedures and assessments plan by fulfilling the Case Report Form (CRF), in the following stages: First visit (Screening); TP - Implants placement; T0 - Implant Loading; TF - final prosthesis T6, T12, T24 and T36 - 6, 12, 24 and 36 months, respectively, after implant loading.

Panoramic radiographs, periapical radiographs, and computed tomography (CT) scans will be obtained from the region of interest before surgery, for surgical planning. Additionally, standardized digital periapical radiographs will be taken in a usual daily practice frequency, as determined by the investigator: after implants placement (TP - immediately or within 1 week after implant placement) and during the post-operative stages (T0, TF, T6, T12, T24, and T36) to assess the osseointegration process, changes in peri-implant bone level as well as prosthetic settlement and integrity.

Moreover, soft tissue evaluation will be conducted at the pre-treatment (Screening visit), for the regions to be rehabilitated with the study implants and in the postoperative period, at T0, TF, T6, T12, T24, and T36, for all study implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years of age or more
* At least one edentulous site in the region of lateral incisors in the maxilla and/or lateral and central incisors in the mandible
* Presence of natural adjacent and opposing tooth,
* Qualified for rehabilitation with narrow implants and single-unit fixed prostheses.

Exclusion Criteria:

As exclusion criteria, the contraindications, and warnings according to the Instructions for Use of the device will be applied, as follows:

* Signs of allergy or hypersensitivity to titanium
* Periodontal disease
* heavy smoking/alcohol drinking habits
* bruxism
* high use of bisphosphonate drugs or proton pump inhibitors (PPIs)
* radiation therapy
* diabetes
* autoimmune diseases
* uncontrolled systemic complications or diseases
* incomplete jawbone growth
* bleeding disorders
* HIV
* osteoporosis
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting 18 years of age or more, with at least one edentulous site in the region of lateral incisors in the maxilla and/or lateral and central incisors in the mandible, who are qualified for rehabilitation with narrow implants and single-unit fixed prostheses.
  Patients that give written informed consent to participate in this clinical study.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Peri-implant bone level change | up to 36 months
  Amount of peri-implant bone level change

SECONDARY OUTCOMES:
Periimplant bone level | up to 36 months
  The peri-implant bone level will be measured on the periapical radiographs obtained as the distance between the coronal margin of the implant shoulder and the most coronal point of the peri-implant bone, on the mesial and distal surfaces of each implant. The horizontal measurement of the remodeling will be done, when there is no bone contact in the cervical part of the implant. This measurement will be performed from the superior site of the bone crest to the lateral edge of the implant, perpendicular to the long axis of the implant.
Implant Survival | up to 36 months
  Implant survival will be defined as the absence of implant loss at each follow-up.
Implant success | up to 36 months
  The implant success will be assessed according to:
  * Absence of persisting subjective discomfort such as pain, foreign body perception, and or dysaesthesia (painful sensation);
  * Absence of recurrent peri-implant infection with suppuration (infection is termed recurrent if observed at two or more follow-up visits after the treatment with systemic antibiotics);
  * Absence of implant mobility on manual palpation;
  * Absence of any continuous peri-implant radiolucency.
Prosthetic Survival | up to 36 months
  Prosthetic survival will be assessed as the final prosthesis remaining in situ at each follow-up, irrespective of its condition.
Prosthetic Success | up to 36 months
  Success will be defined as the prosthesis that remained unchanged and did not require any intervention, except routine occlusal adjustments, during the entire observational period.
Patient Satisfaction with treatment: questionnaire | up to 36 months
  Portuguese translation of the OHIP-14 [20,21] (Annex III) questionnaire will be used to assess Oral Health-Related Quality of Life (OHRQoL), as a measure of patient satisfaction with treatment. Patients will be asked how frequently they have been experiencing the problems assessed by the questionnaire.
Clinician Satisfaction with treatment: questionnaire | up to 36 months
  The assessment will be performed by means of a questionnaire using a visual analog scale (VAS) in the form of a 10 cm horizontal line, where 0 (left end) indicates minimum satisfaction and 10 (right end) indicates maximum satisfaction. The clinician will evaluate his/her satisfaction with the surgical procedure, experience with the use of the abutments, as well as with the surgical and prosthetic results obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Waleska C Furquim, PhD, Study Director — Neodent
Locations (2):
- Brazil (2):
  - Escola de Aperfeiçoamento Profissional dos Cirurgiões Dentistas de Goiás, EAPGOIAS., Goiânia, Goiás
  - Universidade Federal de Uberlândia, Faculdade de Odontologia, Área de Oclusão Prótese Fixa e Materiais Odontológicos., Uberlândia, Minas Gerais

IPD SHARING:
Plan to Share IPD: No